CLINICAL TRIAL: NCT06137690
Title: Factors on Therapeutic Drug Monitoring and Safety of Voriconazole in Critically Ill Elderly Patients: A Prospective Observational Study
Brief Title: Factors on Therapeutic Drug Monitoring and Safety of Voriconazole in Critically Ill Elderly Patients
Status: Recruiting | Type: Observational
Sponsor: People's Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, LIjuan Zhou, Principal Investigator, People's Hospital of Zhengzhou University
Other Study IDs: LJzhou
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Invasive Fungal Infection
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Group A: the elderly group , the age ≥ 60 years
  Interventions: Device: other antifungal agents,breathing machine
- Group B: the non-elderly group , the age < 60 years
  Interventions: Device: other antifungal agents,breathing machine

INTERVENTIONS:
Device: other antifungal agents,breathing machine — If treatment failure for patients in group A and group B，change other antifungal agents (Amphotericin B for Injection, 25mg, North China Pharmaceutical Co., Ltd or Caspofungin Acetate for lnjection,50mg and 70mg Cancidas®). Mechanical ventilation (EVITA 4, Dräger Medical Equipment (Shanghai) Co.,Ltd) was adopte.Treatment failure was defined as no improvement or worse of clinical symptoms, laboratory data, requiring change of antifungal agents therapy.

SUMMARY:
This was a prospective clinical study that all voriconazole-treated adult Chinese patients with invasive pulmonary infection admitted to Zhengzhou Central Hospital affiliated to Zhengzhou University from July 2018 to June 2023. The initial voriconazole serum trough concentration, Correlation of various factors, and risk prediction factors for voriconazole serum trough concentration and hepatotoxicity were compared between elderly and non-elderly patients.

DETAILED DESCRIPTION:
A prospective observational study was conducted from July 2018 to June 2023 in Zhengzhou Central Hospital Affiliated to Zhengzhou University. This study was carried out in accordance with the following criteria: (1) patients who met the criteria for diagnosis of IFI, (2) age ≥ 18 years, (3) The duration of VCZ treatment course ≥ 7 days.

Patients were excluded who fulfilled any of the following criteria: (1) Patients who allergic to VCZ, (2) use other anti-fungal drugs during the use of VCZ, (3) do not qualify for blood sampling monitored by blood concentration, (4) pregnant or lactating women, (5) patients who haven't completely and accurately efficacy and safety data, (6) patients who are treated with a combination of liver enzyme inducers and inhibitors (carbamazepine, phenobarbital, phenytoin, cimetidine, rifampin, rifapentine, rifabutin, and so on),(7) patients who are treated with a combination of Paxlovid or Azvudine.

Grouping: Patients were divided into the elderly group (group A, ≥ 60 years) and the non-elderly group (group B, < 60 years) according to ages. All the recruited patients were treated with voriconazole. Voriconazole was intravenously administered 2 times at the loading dose of 6 mg/Kg or orally administered 2 times at the loading dose of 400mg at 12h intervals, followed by a maintenance dose of 4 mg/Kg or 200 mg at 12 h intervals.

ELIGIBILITY:
Inclusion Criteria:

* patients who met the criteria for diagnosis of IFI
* age ≥ 18 years
* The duration of VCZ treatment course ≥ 7 days.

Exclusion Criteria:

* Patients who allergic to VCZ
* use other anti-fungal drugs during the use of VCZ
* do not qualify for blood sampling monitored by blood concentration
* pregnant or lactating women
* patients who haven't completely and accurately efficacy and safety data
* patients who are treated with a combination of liver enzyme inducers and inhibitors(carbamazepine, phenobarbital, phenytoin, cimetidine, rifampin, rifapentine, rifabutin, and so on)
* patients who are treated with a combination of Paxlovid or Azvudine.

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All voriconazole-treated adult Henan Chinese Han patients with invasive pulmonary infection were admitted to Zhengzhou Central Hospital affiliated to Zhengzhou University from July 2018 to June 2023.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Serum voriconazole trough concentrations | 0.5 hour before voriconazole administration on the Third or sixth day.
  If all patients were administrated by loading dose, voriconazole trough samples were taken immediately 30 minutes before voriconazole administration on the Third day. If all patients were not administrated by loading dose, voriconazole trough samples were taken immediately 30 minutes before voriconazole administration on the sixth day. Blood samples for 2-3 mL were collected in blood-collection tubes without any additives and centrifuged at 3500 rpm for 10min. Serum trough concentrations were determined by a high-performance liquid chromatography method as previously described. A initial steady-state trough concentration blood sample was obtained before dose adjustment for all patients. Each patient received at least one steady-state blood sample. The detections were completed in Translational Medicine Center of Zhengzhou Central Hospital affiliated to Zhengzhou University.
CYP2C19 Genotyping | Unlimited blood drawing time.
  CYP2C19 genotype was determined from peripheral blood, which was extracted and stored in an EDTA anticoagulant tube. Real-time fluorescence quantitative PCR (ThermoFisher Applied Biosystems 7500 fast PCR) was performed using a Human CYP2C19 gene detection kit (PCR-fluorescence probe method, Wuhan YZY Medical Science and Technology Co., Ltd, China) following the manufacturer's instructions. Genomic DNA was isolated from whole blood using QIAamp DNA blood kits (Qiagen, Hilden, Germany). According to nomenclature by the Clinical Pharmacogenetics Implementation Consortium (CPIC®), the CYP2C19 genotype was classified as ultrarapid metabolizer (*17/*17), rapid metabolizer (*1/*17), normal metabolizer (*1/*1), intermediate metabolizer (*1/*2, *1/*3, *2/*17, *3/*17), or poor metabolizer (*2/*2, *2/*3, *3/*3).
The difference of average voriconazole serum trough concentration between group A and group B | From July 2018 to June 2023
  The differences were counted between group A and group B by measuring each patient's voriconazole serum trough concentration.
Analysis of factors affecting voriconazole serum trough concentration | From July 2018 to June 2023
  A multiple linear stepwise regression analysis was performed by using voriconazole serum trough concentration (Y) as the dependent variable, and sex (x1), age (x2), body weight (x3), VCZ route of administration (x4), CYP2C19 phenotype (x5), the average daily dose (x6), PPIs (x7), methylprednisolone (x8), CRP (x9) , PCT (x10), IL-6 (x11), Albumin (x12), ALP (x13), and TBIL (x14) as independent variables. Linear regression analysis reveals the regression equation and independent risk factors affecting voriconazole serum trough concentration.

SECONDARY OUTCOMES:
C-reaction protein (CRP) | Before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy
  It was completed before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy in Zhengzhou city clinical inspection center.
Alanine aminotransferase (ALT) | Before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy
  It was completed before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy in Zhengzhou city clinical inspection center.
Aspartatrtransaminase (AST) | Before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy
  It was completed before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy in Zhengzhou city clinical inspection center.
Gamma-glutamyl transferase(GGT) | Before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy
  It was completed before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy in Zhengzhou city clinical inspection center.
Alkaline phosphatase (ALP) | Before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy
  It was completed before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy in Zhengzhou city clinical inspection center.
Total bilirubin (TBIL) | Before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy
  It was completed before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy in Zhengzhou city clinical inspection center.
procalcitonin(PCT) | Before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy
  It was completed before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy in Zhengzhou city clinical inspection center.
interleukin- 6(IL-6) | before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy
  It was completed before initiation, On the day of blood sample extraction with serum trough concentration, and completion of voriconazole therapy in Zhengzhou city clinical inspection center.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengzhou Central Hospital affiliated to Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No